CLINICAL TRIAL: NCT04423354
Title: A Prospective Clinical Study of Transthoracic Single-hole Assisted Laparoscopic Radical Gastrectomy for Siewert Type Ⅱ Adenocarcinoma of Esophagogastric Junction
Brief Title: A Prospective Clinical Study of Transthoracic Single-hole Assisted Laparoscopic Radical Gastrectomy for Siewert Ⅱ AEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wei Wang, Chief physician, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WWang
Record Dates: First submitted 2020-03-26; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Esophagogastric Junction Adenocarcinoma; Siewert Type II Adenocarcinoma of Esophagogastric Junction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research group (Experimental): Patients diagnosed with Siewert Ⅱ adenocarcinoma of esophagogastric junction and met the inclusion criteria will be assigned to the research group and carry out transthoracic single-hole assisted laparoscopic radical gastrectomy.
  Interventions: Procedure: Transthoracic Single-hole Assisted Laparoscopic Radical Gastrectomy for Siewert Type Ⅱ Adenocarcinoma of Esophagogastric Junction

INTERVENTIONS:
Procedure: Transthoracic Single-hole Assisted Laparoscopic Radical Gastrectomy for Siewert Type Ⅱ Adenocarcinoma of Esophagogastric Junction — Patients diagnosed with Siewert Ⅱ adenocarcinoma of esophagogastric junction and met the inclusion criteria will be assigned to the research group and carry out transthoracic single-hole assisted laparoscopic radical gastrectomy by the fixed surgical group.The same model surgical instruments will be provided by the same instrument company.

SUMMARY:
Objective: To evaluate the safety, feasibility and clinical efficacy of transthoracic single-hole assisted laparoscopic radical gastrectomy for Siewert Type Ⅱ adenocarcinoma of esophagogastric junction.

Methods: A prospective, single-center, one-arm study will be performed. Patients who have been diagnosed with Siewert type Ⅱ esophagogastric junction adenocarcinoma and meet the eligibility criteria will be included in the study and undergo the transthoracic single-hole assisted laparoscopic radical gastrectomy. The data of preoperative, intraoperative, postoperative and follow-up will be recorded and analyzed.

Primary study endpoints: The incidences of early postoperative complications and mortality.

The secondary study endpoints:(1) Surgery and oncology indicators ;(2) Early postoperative recovery information ;(3) 3-year disease-free survival and overall survival rate;(4) 5-year disease-free survival and overall survival.

DETAILED DESCRIPTION:
1. Surgery and oncology indicators,such as length of operation, intraoperative blood loss, transit thoracotomy or laparotomy rate, length of proximal tumor from esophageal resection margin, number of mediastinal lymph node dissections and the positive, number of abdominal lymph node dissections and the positive, tumor type and pathological stage, etc.;
2. Early postoperative recovery information ,such as time of first exhaust and defecation, time of leaving the bed, time of recovery of full and half-flow diet, time of removal of chest drainage tube, time of postoperative hospitalization, etc.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of patients;
* The tumor invaded the anatomy esophagogastric junction (EGJ), with the tumor center located at the EGJ line from 1cm above to 2cm below(SiewertⅡ).
* The endoscopic biopsy was diagnosed with adenocarcinoma;
* Preoperative clinical staging was cT1-4aNanyM0
* No distant metastasis and invasion of surrounding organs were found;
* ECOG score ranged from 0 to 1;
* ASA score ranged from I to III.

Exclusion Criteria:

* Pregnant or lactating women
* Have a severe mental illness
* History of esophagectomy and gastrectomy (including EMR / ESD for gastric and esophageal cancer)
* History of other malignant tumors within 5 years
* History of unstable angina pectoris or myocardial infarction within 6 months
* FEV1% of pulmonary function test was less than 50% of expected value
* History of cerebral infarction or cerebral hemorrhage within 6 months
* Have severe liver and kidney damage

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidences of early perioperative complications | Within 30 days after surgery
  The early perioperative complications include anastomotic fistula, anastomotic stenosis, gastrointestinal dysfunction, chest or abdominal infection, chest or abdominal hemorrhage, respiratory complications, cardiovascular and cerebrovascular accidents, embolism and so on.
Perioperative mortality | Within 30 days after surgery
  The incidence of death due to the surgery

SECONDARY OUTCOMES:
Duration of operation | From the beginning of anesthesia to the completion of surgery
  The time it takes to complete the operation
Intraoperative blood loss | From the beginning of anesthesia to the completion of surgery
  Total blood lost during surgery
The rate of transit thoracotomy or laparotomy | From the beginning of anesthesia to the completion of surgery
  Thoracic or abdominal incisions greater than 10cm are considered to be converted to open chest or abdomen.
Intraoperative mortality | From the beginning of anesthesia to the completion of surgery
  The rate of death during the surgery.
Proximal marginal distance | From the beginning of anesthesia to the completion of surgery
  The length of proximal tumor from esophageal resection margin.
The number of mediastinal lymph node dissections and the positive | About 7 days.
  The mediastinal lymph nodes include NO.19,NO.20,NO.105,NO.106,NO.107,NO.108,NO.109,N0.110,NO.111,NO.112.
The number of abdominal lymph node dissections and the positive | About 7 days.
  The abdominal lymph nodes include NO.1,NO.2,NO.3,NO.4,NO.5,NO.6,NO.7,NO.8,NO.9,NO.10,NO.11,NO.12,NO.13,NO.14.
The tumor type | About 7 days.
  Such as squamous cell carcinoma, adenocarcinoma, etc.
The pathological stage | About 7 days.
  Refer to AJCC 8th Edition TNM staging criteria for esophagus and esophagogastric junction cancer
The duration of first exhaust | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to the first exhaust after the operation.
The duration of first defecation | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to the first defecation after the operation.
The duration of first leaving the bed | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to the first leaving the bed after the operation.
The duration of restoration of full flow diet | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to restore to a full-flow diet after the operation.
The duration of restoration of half-flow diet | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to restore to a half-flow diet after the operation.
The duration of removal of chest drainage tube | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to remove the chest drainage tube after the operation.
The duration of postoperative hospitalization | Time from end of surgery to discharge,about 7 days.
  The duration from the end of the operation to hospital discharge.
3-year overall survival rate | 3 years after surgery
  Overall survival rate during 3 years after surgery
3-year disease-free survival rate | 3 years after surgery
  Disease-free survival rate during 3 years after surgery
5-year overall survival rate | 5 years after surgery
  Overall survival rate during 5 years after surgery
5-year disease-free survival rate | 5 years after surgery
  Disease-free survival rate during 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: wei wang, M.D.,Ph.D, Principal Investigator — Guangdong PHTCM
Locations (1):
- Guangdong Province Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China